CLINICAL TRIAL: NCT03658447
Title: Phase Ib/II Study of Radionuclide 177Lutetium-PSMA-617 Therapy in Combination With Pembrolizumab for Treatment of Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: PRINCE (PSMA-lutetium Radionuclide Therapy and ImmuNotherapy in Prostate CancEr)
Acronym: PRINCE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PeterMac project no. 18/114
Record Dates: First submitted 2018-08-23; First posted 2018-09-05 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-PSMA + Pembrolizumab (Experimental): 200mg pembrolizumab given 3 weekly for upto 35 cycles and 6-weekly 177Lu-PSMA treatments for upto 6 cycles starting at 8.5GBq with administered radioactivity reduced by 0.5GBq for each cycle.
  Interventions: Drug: Pembrolizumab; Drug: 177Lu-PSMA

INTERVENTIONS:
Drug: Pembrolizumab — 200mg Pembrolizumab given 3 weekly for upto 35 cycles
  Other Names: Keytruda
Drug: 177Lu-PSMA — 6-weekly 177Lu-PSMA treatments for upto 6 cycles starting at 8.5GBq with administered radioactivity reduced by 0.5GBq for each cycle.

SUMMARY:
This investigator driven study will examine the safety, tolerability and efficacy of the combination of 177Lutetium-PSMA (177Lu-PSMA) and pembrolizumab in patients with metastatic Castration Resistant Prostate Cancer (mCRPC). 177Lu-PSMA is a compound that binds to the extra-cellular domain of the prostate-specific membrane antigen. Pembrolizumab is an antibody targeted against anti-programmed cell death 1 (PD-1).This is a single arm study where all patients will be treated with 177Lu-PSMA for upto 6 doses and pembrolizumab for upto 35 cycles.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

1. Patient who are at least 18 years of age who have provided written informed consent.
2. Histologically confirmed adenocarcinoma of the prostate without neuroendocrine or small cell differentiation.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 (see Appendix 1).
4. Patients must have progressed on prior enzalutamide, abiraterone and/or apalutamide for treatment of prostate cancer.
5. Determination of disease progression on second generation androgen receptor targeted agent determined by the local investigator. Progressive disease is defined by PCWG3 as any one of the following:

   * PSA progression: minimum of two rising PSA values from a baseline measurement with an interval of ≥ 1 week between each measurement. The PSA value at screening should be ≥ 1ng/ml.
   * Soft tissue or visceral disease progression as per modified RECIST 1.1 criteria (see Appendix 2)
   * Bone progression: ≥ 2 new lesions on bone scan (Appendix 2)
6. At least 2 weeks since the completion of surgery or radiotherapy prior to registration. Any clinically relevant sequelae from the surgery or radiotherapy must have improved to grade 1 prior to registration.
7. Prior surgical orchiectomy or chemical castration maintained on luteinizing hormone-releasing hormone (LHRH) analog (agonist or antagonist). Patients without prior surgical castration must be currently taking and willing to continue luteinizing hormone-releasing hormone (LHRH) analog (agonist or antagonist) therapy throughout the duration of study treatment.
8. Serum testosterone levels ≤ 50ng/dL. (≤ 1.75nmol/L) within 28 days before registration.
9. Imaging evidence of metastatic disease documented with either bone scan or CT scan (Appendix 2).
10. Prior prostate cancer vaccine therapy, radiation therapy, systemic therapies, diethylstilboestrol (DES) or other estrogens are allowed up to 28 days prior to trial registration. Note: bicalutamide flutamide or nilutamide must be discontinued within 4 weeks of registration.
11. Significant PSMA avidity on 68Ga/18F-PSMA PET/CT, defined as a minimum uptake of SUVmax 20 at a site of disease, and SUVmax > 10 at other sites of disease ≥10mm (unless subject to factors explaining a lower uptake, e.g. respiratory motion, reconstruction artefact).
12. Patients must have a life expectancy ≥ 24 weeks.
13. Patients must agree to use a highly effective form of contraception for the entire duration of the study plus an additional 120 days (a spermatogenesis cycle) after the last dose of study treatment and refrain from donating sperm during this period (see section 10.3.3).
14. Patients must be willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled assessments.
15. Patients must have adequate bone marrow, hepatic and renal function documented within 28 days of registration, defined as:

    * Haemoglobin ≥90 g/L independent of transfusions (no red blood cell transfusion in last 4 weeks)
    * White blood cells >3x109/L
    * Absolute neutrophil count ≥1.5x109/L
    * Platelets ≥100 x109/L
    * Total bilirubin ≤1.5 x upper limit of normal (ULN) except for patients with known Gilbert's syndrome.
    * Aspartate transaminase (AST) (SGOT) and alanine transaminase (ALT) (SGPT) ≤2.5 × ULN or ≤5 × ULN for participants with liver metastases.
    * Serum creatinine ≤1.5 x ULN or a calculated creatinine clearance > 50mL/min (Chronic Kidney Disease Epidemiology (CKD-EPI) equation for patients with creatinine levels above institutional normal.
    * Albumin >30 g/dl
    * International normalized ratio (INR), prothrombin time (PT), activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
16. Patients who are deemed by PSMA imaging to have readily accessible disease will be required to consent to 3 serial tumour biopsies - at screening, post combination treatment (at any time between weeks 2-4) and on progression

Exclusion Criteria:

1. Site(s) of disease that are FDG positive with low PSMA expression defined by PSMA SUVmax < 10.
2. Previous history or presence of brain metastases or leptomeningeal metastases.
3. Any prior exposure to anti-PD-1, anti-PD-L1/L2, anti-CTLA-4 antibody or any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathway.
4. Any prior treatment with cabazitaxel.
5. Any prior exposure to 177Lu-PSMA.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Patients with active, known or suspected autoimmune disease including Sjogren's syndrome. Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are eligible.
8. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
9. Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy may be eligible.
10. Patients with a condition requiring systemic treatment with either corticosteroids (> 10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of registration. Inhaled or topical steroids, and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
11. Other malignancies within the previous 2-years other than, melanoma in situ, basal cell or squamous cell carcinomas of skin with a > 30% probability of recurrence within 12 months.
12. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
13. Patient has a known history of Human Immunodeficiency Virus (HIV).
14. Patients with symptomatic or impending cord compression unless appropriately treated beforehand and clinically stable for ≥ 4 weeks.
15. Previous history of interstitial lung disease or non-infectious pneumonitis.
16. Recent administration of a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
17. Recent administration of the influenza vaccine (within 30 days of registration).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with mCRPC who are minimally symptomatic and have progressed on at least one line of novel AR targeted agents (e.g. enzalutamide, abiraterone acetate, apalutamide, etc.) will be eligible for the study. Patients may have received docetaxel chemotherapy in the treatment naïve or castrate resistant setting. Patients already receiving anti-bone resorptive therapy for management of SREs are permitted to continue with this treatment.
Enrollment: 37 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Prostate Specific Antigen (PSA) response | Through study completion, up until 24 months after the last patient commences treatment.
  PSA response will be defined as a 50% or greater decrease in PSA from baseline to the lowest post-baseline PSA result. A second consecutive value obtained 3 or more weeks later is required to confirm the PSA response.
Incidence of Treatment-Emergent Adverse Events [Safety] | Through treatment completion, maximum of 24 months
  Safety will be measured by serious adverse events (SAEs) and AEs assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Tolerability | Through treatment completion, maximum of 24 months
  Tolerability is defined as the time from treatment commencement until treatment discontinuation due to toxicity. Participants who ceased treatment due to reasons other than toxicity will be censored at the time of ceasing protocol treatment and participants who died while on treatment from reasons unrelated to the treatment will be censored at the date of death.

SECONDARY OUTCOMES:
Radiographic progression free survival | Through study completion, up until 24 months after the last patient commences treatment.
PSA-progression free survival | Through study completion, up until 24 months after the last patient commences treatment.
  Time from treatment initiation to the date of PSA progression per PCWG3 or death due to any cause, whichever occurs first. The date of PSA progression is the date that an increase of 25% or more and an absolute increase of 2ng/mL or more from the nadir is documented.
Overall survival | Through study completion, up until 24 months after the last patient commences treatment
Overall Response Rate by modified RECIST1.1 | Through study completion, up until 24 months after the last patient commences treatment
Duration of objective tumour response as assessed by modified RECIST 1.1 for soft tissue and PCWG3 for bone lesions | Through study completion, up until 24 months after the last patient commences treatment
Time to treatment (TTR) response | Through study completion, up until 24 months after the last patient commences treatment
  TTR-PCWG3 is defined as the time from treatment initiation to the date of the first documented CR or PR per modified RECIST1.1 for soft tissue and PCWG3 for bone lesions.
Change in pain | Through treatment completion, maximum of 24 months
  The Brief Pain Inventory - Short Form (BPI-SF) is 15-item domain-specific instrument designed to assess the severity of pain and the impact/interference of pain on daily functions through the use of a numerical rating scale (NRS). Participants rate the severity of their pain as its "worse", "least' and "average" in the last 24 hours using an 11-point NRS with anchors "no pain'' and ''pain as bad as you can imagine.'' This instrument consists of 2 domains: pain severity and pain interference. The BPI-SF also asks the participants to mark the location of the pain on a body drawing and includes additional questions regarding pain treatment and the extent of pain relief. The BPI-SF will be scored according to the user guide. Higher pain scores is worse outcome.
Change in Health Related Quality of Life (HRQoL) | Through treatment completion, maximum of 24 months
  The Functional Assessment of Cancer Therapy - Prostate cancer (FACT-P) provides information about general and disease-specific symptoms. The FACT-P module is a disease-specific 39-item questionnaire that has been validated for the purpose of assessing health-related quality of life (HRQoL) in prostate cancer patients. The FACT-P consists of 5 subscales: Physical Well-Being (7 items), Functional Well-Being (7 items), Emotional Well-Being (6 items), Social Well- Being (7 items), and additional concerns or Prostate Cancer Subscale (PCS) specific to prostate cancer (12 items). FACT-P questions are scored on a 5-point Likert scale from 0 to 4 (0 being not at all and 4 being very much).Scoring of the FACT-P will be based on the user manual. Higher scores means higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Shahneen Sandhu, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (4):
- Australia (4):
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No